CLINICAL TRIAL: NCT06750458
Title: Comparative Study Between Dapagliflozin Versus Dexamethasone Role in Pre-operative Management of Non- Diabetic Brain Tumor Patients
Brief Title: Dapagliflozin Versus Dexamethasone Role in Pre-operative Management of Non- Diabetic Brain Tumor Patients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Maha Khalifa, PhD Candidate, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 36265MD324/12/24
Record Dates: First submitted 2024-12-15; First posted 2024-12-27 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Glioma; Dapagliflozin (Forxiga); Dexamethasone
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- GroupⅠ(n=25) (Control group) (Placebo Comparator): This group will include twenty-five non-diabetic glioma patients on levetiracetam, and not on SGLT2 inhibitors who will receive placebo tablets once daily for 14 days pre-operative.
  Interventions: Drug: Placebo
- GroupII (n=25) (Dapagliflozin group) (Experimental): This group will include twenty-five non-diabetic glioma patients on levetiracetam, and not on SGLT2 inhibitors who will receive Dapagliflozin 10 mg once daily for 14 days pre-operative.
  Interventions: Drug: Dapagliflozin placebo
- Group III (n=25) (Dexamethasone group)This group will include twenty-five non-diabetic glioma patien (Active Comparator): This group will include twenty-five non-diabetic glioma patients on levetiracetam, and not on SGLT2 inhibitors who will receive Dexamethasone 8 mg tablets once daily for 14 days pre-operative.
  Interventions: Drug: DexamethasoneGroup III (n=25) (Dexamethasone group)

INTERVENTIONS:
Drug: Dapagliflozin placebo — Twenty-five non-diabetic glioma patients on levetiracetam, and not on SGLT2 inhibitors will receive Dapagliflozin 10 mg once daily for 14 days pre-operative
  Arms: GroupII (n=25) (Dapagliflozin group)
Drug: Placebo — Twenty-five non-diabetic glioma patients on levetiracetam, and not on SGLT2 inhibitors will receive placebo tablets once daily for 14 days pre-operative.
  Arms: GroupⅠ(n=25) (Control group)
Drug: DexamethasoneGroup III (n=25) (Dexamethasone group) — Twenty-five non-diabetic glioma patients on levetiracetam, and not on SGLT2 inhibitors will receive Dexamethasone 8 mg tablets once daily for 14 days pre-operative.
  Arms: Group III (n=25) (Dexamethasone group)This group will include twenty-five non-diabetic glioma patien

SUMMARY:
The aim of the study is to compare between the role of dapagliflozin versus dexamethasone in pre-operative management of non-diabetic glioma patients on levetiracetam as anti-seizure drug.

DETAILED DESCRIPTION:
* This is a randomized, parallel, and controlled study, which will be conducted on pre-operative non-diabetic glioma patients on levetiracetam as anti-seizure drug. * This study will be conducted pending registration at ClinicalTrials.gov.
* All patients will give their written informed consents.
* Data of patients will be confidential.
* Any unexpected risk will be reported to patients and Ethical Committee on time. * Randomization will be carried out based on days on hospital admission.

ELIGIBILITY:
Inclusion Criteria:

* Males & females.
* Age: between 18 and 75 years old.
* Pre-operative non-diabetic glioma patients on levetiracetam. • Diagnosis will be confirmed by:

  * The initial clinical examination.
  * Magnetic resonance imaging of the brain (MRI) with contrast.

Exclusion Criteria:

* Age: > 75 years old, and <18 years old.
* Breast feeding female. • Pregnant female.
* eGFR< 30 mL/minute/1.73 m2.
* Patients with diabetes mellitus.
* Patients with diabetic ketoacidosis.
* Patients with urinary tract infection.
* Dehydrated patients till normalized.
* Lower limb amputation patients.
* SGLT2 inhibitors hypersensitivity.
* Severe hepatic patients (child-plug score class-c).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2026-10-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
•Magnetic resonance imaging of the brain (MRI) with contrast. | 2 weeks
Optic nerve sheath diameter for assessment of intracranial tension. | 2 weeks

SECONDARY OUTCOMES:
Tumor necrosis factor alpha (TNF-α). | 2 weeks
Interlukin-6 (IL-6). | 2 weeks

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Takashima M, Nakamura K, Kiyohara T, Wakisaka Y, Hidaka M, Takaki H, Yamanaka K, Shibahara T, Wakisaka M, Ago T, Kitazono T. Low-dose sodium-glucose cotransporter 2 inhibitor ameliorates ischemic brain injury in mice through pericyte protection without glucose-lowering effects. Commun Biol. 2022 Jul 2;5(1):653. doi: 10.1038/s42003-022-03605-4. PMID 35780235
- [Result] Shim B, Stokum JA, Moyer M, Tsymbalyuk N, Tsymbalyuk O, Keledjian K, Ivanova S, Tosun C, Gerzanich V, Simard JM. Canagliflozin, an Inhibitor of the Na+-Coupled D-Glucose Cotransporter, SGLT2, Inhibits Astrocyte Swelling and Brain Swelling in Cerebral Ischemia. Cells. 2023 Sep 6;12(18):2221. doi: 10.3390/cells12182221. PMID 37759444
- [Result] Saeedi S, Rezayi S, Keshavarz H, R Niakan Kalhori S. MRI-based brain tumor detection using convolutional deep learning methods and chosen machine learning techniques. BMC Med Inform Decis Mak. 2023 Jan 23;23(1):16. doi: 10.1186/s12911-023-02114-6. PMID 36691030
- [Result] Weller M, Wen PY, Chang SM, Dirven L, Lim M, Monje M, Reifenberger G. Glioma. Nat Rev Dis Primers. 2024 May 9;10(1):33. doi: 10.1038/s41572-024-00516-y. PMID 38724526